CLINICAL TRIAL: NCT02110810
Title: Rectal Indomethacin Decreases the Incidence of Pancreatitis Following Endoscopic Retrograde Cholangiopancreatography in High-risk Patients
Brief Title: Indomethacin Decreases Post-ERCP Pancreatitis
Acronym: Indomethacin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Alejandro Gonzalez-Ojeda, PhD. MD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Indomethacin-2014-02
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Post ERCP Acute Pancreatitis
Keywords: post-ERCP Acute Pancreatitis; Indomethacin; NSAIDs
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin (Experimental): 100 mg of Indomethacin suppository immediately afterwards while still under sedation
  Interventions: Drug: Indomethacin
- 2.6-g suppository of glycerin (Placebo Comparator): suppository of 2.4 g of glycerin immediately afterwards while still under sedation
  Interventions: Drug: 2.6-g suppository of glycerin

INTERVENTIONS:
Drug: Indomethacin — Indomethacin suppository of 100 mg immediately afterwards while still under sedation
  Arms: Indomethacin
Drug: 2.6-g suppository of glycerin — to receive a 2.4 g of glycerin suppository immediately afterwards while still under sedation
  Other Names: glycerin suppository
  Arms: 2.6-g suppository of glycerin

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is now a widely accepted therapy for treating benign and malignant diseases of the pancreatobiliary tree. Acute pancreatitis represents the most common and feared complication following ERCP. The reported incidence of this complication is from 1% to 40% according to the presence of high-risk factors for this complication or the presence dysfunction in the sphincter of Oddi (SOD). In most prospective series, the incidence has ranged between 3.5% and 20% for nonselected and high-risk patients, respectively. Independent risk factors for post-ERCP pancreatitis are either patient- or procedure-related.

DETAILED DESCRIPTION:
Design This is a randomized clinical trial carried out in patients scheduled for ERCP at the Department of Gastrointestinal Endoscopy and Department of Gastroenterology of the Specialties Hospital of the Western Medical Center, in Guadalajara, Jalisco, Mexico. The investigators include patients with an elevated baseline risk of post-ERCP pancreatitis based on prospectively validated patient- and procedure-related independent risk factors.

The ERCP procedures are performed with the patient under topical pharyngeal anesthesia with 2% lidocaine and after administration of sedation (midazolam) and analgesia (fentanyl) intravenously, with dosages at the discretion of the endoscopist. Patients receive complementary oxygen through an external nasal device at 3 to 5 L/min and infusion of 200 to 500 mL of 0.9% sterile saline solution.

The equipment and protocol that are being used to perform ERCP consist of a video duodenoscope (Olympus, Tokyo, Japan), sphincterotome traction for selective cannulation of the bile duct, a needle scalpel to perform precut sphincterotomy, a hydrophilic guide wire via the bile duct, a Dormia basket and/or balloon catheter for stone extraction, and nonionic water-soluble contrast medium at 300 mg/mL (Optira 300™; ioversol injection 64%; Mallinckrodt Pharmaceuticals, Dublin, Ireland) for opacification of the biliary and pancreatic ducts.

Pancreatic stents are being used only to treat pancreatic fistulas and to prevent pancreatitis. All patients are monitored continuously during the procedure, with determinations of blood pressure, heart rate, respiratory rate, and arterial blood oxygen saturation.

Eligible patients who provide written informed consent undergo the randomization at conclusion of the ERCP procedure because patients without risk factors could be included in the study based on procedure-related factors alone. If patients met the inclusion criteria, they are randomly assigned to receive a 100 mg suppository of indomethacin or 2.4 g of glycerin suppository immediately afterwards while still under sedation. All patients are observed to prevent spontaneous expulsion of the suppository until they became completely awake. All patients, staff endoscopists, residents, and researchers are blinded to the treatment assigned to each of them.

The following data that is being collected.

1. A clinical history, particularly patient-related risk factors for post-ERCP pancreatitis; blood test results for the determination of basal amylase, liver enzymes, and bilirubin levels; as well as results of ultrasonography of the liver and biliary tract.
2. All data generated during the ERCP is being recorded, particularly those related to procedure-related risk factors for developing acute pancreatitis. In addition, other nonpancreas-related complications are being recorded as perforation or bleeding.
3. Any adverse events related to the rectally applied indomethacin or glycerin suppositories are being recorded as expulsion, irritation, or bleeding.

Post-ERCP pancreatitis is considered the main outcome variable and is defined as the development of new or increased abdominal pain consistent with pancreatitis, and elevated blood amylase or lipase >3 times the upper limit of normal until 24 h after the procedure, and hospitalization (or prolongation of existing hospitalization) for at least 2 nights. The severity is determined according to consensus guidelines, with mild post-ERCP pancreatitis resulting in hospitalization of less than 3 days, and moderate post-ERCP pancreatitis resulting in hospitalization of 4-10 days. Severe post-ERCP pancreatitis is qualified as resulting in a hospitalization of >10 days, or leading to the development of pancreatic necrosis or pseudocysts, or requiring percutaneous or surgical intervention. Patients with acute pancreatitis are being followed up for 30 days after hospital discharge. Asymptomatic hyperamylasemia is defined as any amylase level at least three times above the normal serum level in the absence of abdominal pain.

Follow up The patients are kept under surveillance in the endoscopy recovery area for 3 h after ERCP. Measurement of serum amylase is determined at 2 h post-ERCP in all included patients. Asymptomatic outpatients are discharged after 6 h of surveillance with monitoring for signs and symptoms of acute post-ERCP pancreatitis by telephone contact for 24 hours.

Hospitalized asymptomatic patients are being discharged to their assigned bed after 4 hours of surveillance, where clinical surveillance is continued for up to 24 h. If new abdominal pain suggestive of pancreatic origin appeares at any time, the 2-h amylase level is checked and confirmed with serum lipase determination.

All routine laboratory examinations are being performed when acute pancreatitis of any etiology is established. All patients diagnosed with post-ERCP pancreatitis are being managed under the medical care of the Department of Gastroenterology.

Patients are being submitted to computed tomography scanning to determine the severity of the episode of pancreatitis. Severity was established according to Cotton's criteria.

Statistical analysis Statistical software, SPSS for IBM (version 20 for Windows; IBM Corp., Armonk, NY, USA) is beign used for data analysis.

The data obtained will be expressed as frequencies and percentages, means and standard deviations. For comparing results, Student's t test will be used for continuous variables and Chi2 or Fisher's exact tests will be used for qualitative data when appropriate.

Relative risk (RR) and 95% confidence intervals (95% CI) will be determined as well as the absolute risk reduction (ARR), relative risk reduction (RRR), and number needed to treat (NNT).

Statistical significance from two-tailed tests was assumed when p < 0.05

ELIGIBILITY:
Inclusion Criteria:

* If they met one or more of the following criteria:

  * a clinical suspicion of SOD dysfunction;
  * or a history of post-ERCP pancreatitis, pancreatic
  * or precut sphincterotomy,
  * more than eight cannulation attempts,
  * pneumatic dilatation of an intact biliary sphincter,
  * or ampullectomy
* Patients were also eligible for inclusion if they met two of the following criteria:

  * aged 50 years or younger and female gender
  * or a history of recurrent pancreatitis (>2 episodes),
  * three or more injections of contrast agent into the pancreatic duct with at least one injection to the tail of the pancreas,
  * excessive injection of contrast agent into the pancreatic duct resulting in opacification of pancreatic acini,
  * or the need for acquisition of a cytology specimen from the pancreatic duct with the use of a tissue-sampling brush.

Exclusion Criteria:

* unwillingness or inability to consent for the study
* pregnancy
* breast feeding
* standard contraindications for ERCP
* hypersensitivity to aspirin or NSAIDs
* previous use of NSAIDs within 1 week
* renal failure (creatinine clearance rate >1.4 mg/dL)
* active or recent (< 4 weeks) gastrointestinal hemorrhage
* chronic calcified pancreatitis
* pancreatic head malignancy
* any procedure performed on the major papilla/ventral pancreatic duct in patients with a pancreatic divisum
* previous ERCP for biliary stent removal or exchange without an anticipated pancreatogram
* subjects with prior biliary sphincterotomy and scheduled for repeat biliary therapy without an anticipated pancreatogram
* or anticipated inability to follow our protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Post ERCP Acute Pancreatitis | 48 hours after the procedure.
  Defined as the development of new or increased abdominal pain consistent with pancreatitis, and elevated blood amylase or lipase >3 times the upper limit of normal until 24 h after the procedure, and hospitalization (or prolongation of existing hospitalization) for at least 2 nights.

SECONDARY OUTCOMES:
Severity of post-ERCP pancreatitis | 48 hours after procedure.
  was determined according to consensus guidelines, with mild post-ERCP pancreatitis resulting in hospitalization of < 3 days, and moderate post-ERCP pancreatitis resulting in hospitalization of 4-10 days
Acute Pancreatitis | During 30 days after hospital discharge.
  Patients who developed Acute Pancreatitis after hospital discharge with presence of abdominal pain consistent with pancreatitis, and elevated blood amylase or lipase >3 times the upper limit of normal.
Asymptomatic hyperamylasemia | 48 hours after procedue.
  any amylase level at least three times above the normal serum level in the absence of abdominal pain.
Measurement of serum amylase | 2 hours post-ERCP
  measured in all patients right after procedure and during surveillance (3 hours).
Routine laboratory examinations | 2 hours after procedure and daily until hospital discharge, an expected average of 10 days.
  All laboratory exams were performed when acute pancreatitis of any etiology was established

CONTACTS AND LOCATIONS:
Overall Officials: González-Ojeda Alejandro, Ph.D., M.D., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Department of Gastrointestinal Endoscopy and Department of Gastroenterology of the Specialties Hospital of the Western Medical Center of the Mexican Institute of Social Security., Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Andrade-Davila VF, Chavez-Tostado M, Davalos-Cobian C, Garcia-Correa J, Montano-Loza A, Fuentes-Orozco C, Macias-Amezcua MD, Garcia-Renteria J, Rendon-Felix J, Cortes-Lares JA, Ambriz-Gonzalez G, Cortes-Flores AO, Alvarez-Villasenor Adel S, Gonzalez-Ojeda A. Rectal indomethacin versus placebo to reduce the incidence of pancreatitis after endoscopic retrograde cholangiopancreatography: results of a controlled clinical trial. BMC Gastroenterol. 2015 Jul 21;15:85. doi: 10.1186/s12876-015-0314-2. PMID 26195123